CLINICAL TRIAL: NCT03275402
Title: A Multicenter Phase 2/3 Trial of the Efficacy and Safety of Intracerebroventricular Radioimmunotherapy Using 131I-omburtamab for Neuroblastoma Central Nervous System/Leptomeningeal Metastases
Brief Title: 131I-omburtamab Radioimmunotherapy for Neuroblastoma Central Nervous System/Leptomeningeal Metastases
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Corporate business decision. Not due to safety or efficacy concerns.
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2017-09-06; First posted 2017-09-07 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Neuroblastoma; CNS Metastases; Leptomeningeal Metastases
Keywords: Radioimmunotherapy; Neuroblastoma; CNS Metastases; Leptomeningeal Metastases; Pediatric
MeSH Terms: conditions — Neuroblastoma; Meningeal Carcinomatosis | interventions — omburtamab I-131

STUDY DESIGN:
Intervention Model Description: Patients will receive up to two cycles of intracerebroventricular 131I-omburtamab. Safety and efficacy will be investigated with short-term follow-up at 26 weeks after treatment and with long-term follow-up for up to 3 years following treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 131I-omburtamab (Experimental): One treatment cycle of 131I-omburtamab consists of one dosimetry dose (2 mCi ) (for subjects enrolled on Version 1-7 of Protocol 101) and one treatment dose (50 mCi) for up to 2 cycles of length 5 weeks (for subjects enrolled on Version 1-7 of Protocol 101) or 4 weeks (for subject enrolled after Version 7 of Protocol 101). For Japan only, the first cycle consisted of one dosimetry dose (2 mCi ) week 1 one treatment dose (50 mCi) week 2. If eligible a second cycle of 50 mCi 131I-omburtamab was given at week 6. For subjects below 3 and 1 years of age, the treatment dose was reduced by 33% and 50%, respectively.
  Interventions: Biological: 131I-omburtamab

INTERVENTIONS:
Biological: 131I-omburtamab — Murine IgG1 monoclonal antibody radiolabeled with iodine-131
  Other Names: 131I-8H9

SUMMARY:
Children with a neuroblastoma diagnose and central nervous system (CNS)/leptomeningeal metastases will be given up to 2 rounds of intracerebroventricular treatment with a radiolabelled monoclonal antibody, 131I-omburtamab to evaluate efficacy and safety

DETAILED DESCRIPTION:
One 131I-omburtamab treatment cycle takes 4 weeks and includes a treatment dose, and an observation period and post-treatment evaluations.

One 131I-omburtamab treatment cycle for Japan only takes 5 weeks and includes a dosimetry dose (2mCi) of 131I-omburtamab is administered during week 1 followed by blood/cerebral spinal fluid (CSF) samples and whole-body scintigraphy at predefined intervals during the following 48 hours after treatment.

* A therapeutic dose (50mCi) of 131I-omburtamab is administered during week 1 (week 2 for Japan) followed by a 3-week observation period that includes a repeated MRI, CSF cytology, and safety monitoring.
* A second treatment cycle of 131I-omburtamab is administered during week 5 (week 6 for Japan) if there is no objective disease progression week 5 after the first injection, and the participant is presenting without unexpected and clinical significant Grade 4 toxicity. For participants with ongoing Grade 3 toxicity a second doing cycle will take place according to the discretion of the investigator.

Participants can be treated in an outpatient setting or may be admitted as inpatients for both the dosimetry and the therapeutic injections.

Participants completing at least one treatment period will first enter a follow-up period through week 26 and thereafter the long-term follow-up where patients will be evaluated for up to 3 years post-131I-omburtamab treatment where after the trial is ended

Participants will be monitored for adverse events during and after 131I-omburtamab injection and will have pre- and post-treatment clinical assessments including neurologic examination, hematology and serum chemistry, blood and CSF cultures, endocrinology assessments, CSF analysis, and, pre- and post 131I-omburtamab performance testing. Performance testing will be performed at trial baseline, at week 26 and every 6 months during trial period.

In case the patient has a subsequent relapse in the CNS/LM after 131I-omburtamab therapy during the follow-up period, re-treatment to target minimal residual disease can be considered and allowed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of neuroblastoma with relapse in the central nervous system or in the meninges (leptomeningeal).
* Patients must be between the ages of birth and 18 years at the time of screening.
* Patients must have a life expectancy of at least 3 months.

Exclusion Criteria:

* Patients with primary neuroblastoma in central nervous system.
* Patients must not have an uncontrolled life-threatening infection.
* Patients must not have received cranial or spinal irradiation less than 3 weeks prior to first dose of 131I-omburtamab in this trial.
* Patients must not have received systemic chemotherapy (corticosteroids not included) less than 3 weeks prior to enrollment in this trial.
* Patients must not have severe major non-hematologic organ toxicity; specifically, any renal, cardiac, hepatic, pulmonary, and gastrointestinal system toxicity must fall below Grade 3 prior to enrollment in this trial. Patients with stable neurological deficits (due to brain tumor) are not excluded. Patients with Grade 3 or lower hearing loss are not excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Roemer, MD, Study Director — Y-mAbs Therapeutics
Locations (8):
- United States (5):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Riley Hospital for Children, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
- Rigshospitalet, Copenhagen, Denmark
- Department of Pediatric Oncology Fukushima Medical University Hospita, Fukushima, Japan
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prasad K, Serencsits BE, Chu BP, Dauer LT, Donzelli M, Basu E, Kramer K, Pandit-Taskar N. Feasibility of safe outpatient treatment in pediatric patients following intraventricular radioimmunotherapy with 131I-omburtamab for leptomeningeal disease. EJNMMI Res. 2024 Jul 31;14(1):70. doi: 10.1186/s13550-024-01127-0. PMID 39083105
- [Derived] Prasad K, Serencsits BE, Chu BP, Dauer LT, Donzelli M, Basu E, Kramer K, Pandit-Taskar N. Feasibility of safe outpatient treatment in pediatric patients following intraventricular radioimmunotherapy with 131I-omburtamab for leptomeningeal disease. Res Sq [Preprint]. 2024 Feb 28:rs.3.rs-3969388. doi: 10.21203/rs.3.rs-3969388/v1. PMID 38464207

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 131I-omburtamab
Started | 52
Completed | 13
Not Completed | 39
Not completed — Death | 17
Not completed — Study terminated by sponsor | 21
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- 131I-omburtamab: One treatment cycle of 131I-omburtamab consists of 1 dose at 50mCi at week 1. For Japan only one treatment cycle of 131I-omburtamab consists of 2 doses: 2mCi at week 1 and 50mCi at week 2. First cycle is initiated right after confirmation of eligibility at week 1. At week 5 (week 6 for Japan) the participant will be evaluated for safety and if eligible, receive a second cycle of 131I-omburtamab.
  Secondary efficacy endpoints will be evaluated at week 26 and primary efficacy endpoint will be evaluated at week 156.
  131I-omburtamab: Murine IgG1 monoclonal antibody radiolabeled with iodine-131
Arm/Group | 131I-omburtamab
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (2.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 36
  Japan | 3
  Denmark | 1
  Spain | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate
Description: Overall survival rate at 3 years after the first treatment dose of 131I-omburtamab estimated by the Kaplan-Meier method.
Time Frame: 3 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | 131I-omburtamab
Number analyzed (Participants) | 52
Proportion of participants | 0.65 [0.49 to 0.78]

ADVERSE EVENTS:
Time Frame: Adverse events, including serious, were reported from 1st dose until 3 weeks after the last IMP administration. From 3 weeks after the last IMP administration up to 3 years only SAEs considered related to IMP and new onset for cancers were assessed All cause mortality was assessed up to 3 years.
Description: All adverse events, including serious, were reported from 1st dose until 3 weeks after the last IMP administration. All SAEs were reported. Note that from 3 weeks after last IMP administration and during the 3-year long term follow-up only SAEs considered related to IMP and new onset for cancers were collected.
Arm/Group | 131I-omburtamab
All-Cause Mortality (participants affected / at risk) | 17/52
Serious Adverse Events (participants affected / at risk) | 20/52
Other Adverse Events (participants affected / at risk) | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 131I-omburtamab (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Meningitis chemical (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 8 (9)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 4 (4)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 131I-omburtamab (N=52)
Anaemia (Blood and lymphatic system disorders) | 15 (22)
Tachycardia (Cardiac disorders) | 4 (10)
Hypothyroidism (Endocrine disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 19 (21)
Vomiting (Gastrointestinal disorders) | 18 (25)
Fatigue (General disorders) | 4 (4)
Pain (General disorders) | 6 (20)
Pyrexia (General disorders) | 8 (9)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 16 (19)
Neutrophil count decreased (Investigations) | 22 (43)
Platelet count decreased (Investigations) | 22 (26)
Protein total decreased (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 23 (34)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Headache (Nervous system disorders) | 12 (20)
Neuralgia (Nervous system disorders) | 5 (10)
Irritability (Psychiatric disorders) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (7)
Haematoma (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 4 (8)
Hypotension (Vascular disorders) | 4 (9)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to a business strategy decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03275402/Prot_SAP_000.pdf